CLINICAL TRIAL: NCT02757716
Title: Addiction Remission and Addiction Transfer After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, Dr. med. Sonja Chiappetta, Dr. med. Christine Stier, Sana Klinikum Offenbach
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FF 146/2015
Record Dates: First submitted 2016-04-21; First posted 2016-05-02 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: addiction remission; addiction transfer
MeSH Terms: conditions — Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sleeve Gastrectomy (Other): Obese patients who undergo sleeve gastrectomy fill in questionnaire
  Interventions: Other: Questionnaire
- Roux-en-Y-Gastric Bypass (Other): Obese patients who undergo roux-en-y-gastric bypass fill in questionnaire
  Interventions: Other: Questionnaire
- One anastomosis-Gastric Bypass (Other): Obese patients who undergo one anastomosis gastric bypass fill in questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Every patient who undergo surgery will fill out a questionnaire containing validated scales concerning food, alcohol, nicotine, internet and exercise and drug addiction prior, 6 months and 24 months after surgery.

SUMMARY:
To evaluate addiction remission and addiction transfer after bariatric surgery.

DETAILED DESCRIPTION:
A prospective study to evaluate addiction remission and addiction transfer 6 and 24 months after primary surgery (sleeve gastrectomy, Roux-en-Y- gastric bypass and One anastomosis gastric bypass) in obese patients. A questionnaire evaluating food addiction (Yale Food Scale), alcohol addiction (Audit Scale), nicotine addiction (Fagerström Scale), exercise addiction (Exercise Addiction Inventory), internet addiction (ISS20) and drug addiction (Drug Use Questionnaire) gets completed prior to surgery and 6 and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35kg/m² and obesity related disease or BMI > 40kg/m²

Exclusion Criteria:

* decline of study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Addiction remission | 24 months after surgery
  Addiction remission (evaluated by questionnaire) after obesity surgery

SECONDARY OUTCOMES:
Addiction transfer | 24 months after surgery
  Addiction transfer (evaluated by questionnaire) after obesity surgery
Excess Weight Loss (EWL in %) | 24 months after surgery
  EWL 24 months after surgery measured as a physiological parameter at 2 year Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Weiner, Prof., Study Chair — Sana Klinikum Offenbach, Department of Obesity and Metabolic Surgery
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Offenbach Am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Volkow ND, Wang GJ, Tomasi D, Baler RD. The addictive dimensionality of obesity. Biol Psychiatry. 2013 May 1;73(9):811-8. doi: 10.1016/j.biopsych.2012.12.020. Epub 2013 Jan 29. PMID 23374642
- [Result] Pepino MY, Stein RI, Eagon JC, Klein S. Bariatric surgery-induced weight loss causes remission of food addiction in extreme obesity. Obesity (Silver Spring). 2014 Aug;22(8):1792-8. doi: 10.1002/oby.20797. Epub 2014 May 23. PMID 24852693
- [Result] Cuellar-Barboza AB, Frye MA, Grothe K, Prieto ML, Schneekloth TD, Loukianova LL, Hall-Flavin DK, Clark MM, Karpyak VM, Miller JD, Abulseoud OA. Change in consumption patterns for treatment-seeking patients with alcohol use disorder post-bariatric surgery. J Psychosom Res. 2015 Mar;78(3):199-204. doi: 10.1016/j.jpsychores.2014.06.019. Epub 2014 Sep 7. PMID 25258356
- [Result] Fowler L, Ivezaj V, Saules KK. Problematic intake of high-sugar/low-fat and high glycemic index foods by bariatric patients is associated with development of post-surgical new onset substance use disorders. Eat Behav. 2014 Aug;15(3):505-8. doi: 10.1016/j.eatbeh.2014.06.009. Epub 2014 Jun 20. PMID 25064307
- [Result] Ivezaj V, Saules KK, Wiedemann AA. "I didn't see this coming.": why are postbariatric patients in substance abuse treatment? Patients' perceptions of etiology and future recommendations. Obes Surg. 2012 Aug;22(8):1308-14. doi: 10.1007/s11695-012-0668-2. PMID 22661046
- [Derived] Chiappetta S, Stier C, Hadid MA, Malo N, Theodoridou S, Weiner R, Weiner S. Remission of Food Addiction Does Not Induce Cross-Addiction after Sleeve Gastrectomy and Gastric Bypass: A Prospective Cohort Study. Obes Facts. 2020;13(3):307-320. doi: 10.1159/000506838. Epub 2020 May 5. PMID 32369811